CLINICAL TRIAL: NCT07208721
Title: The Key to Emotional Balance: The Effect of a Positive Psychotherapy-Based Balance Model on Emotion Regulation, Recovery, and Life Purpose in Bipolar Disorder
Brief Title: The Key to Emotional Balance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Eda Albayrak Günday, Research Assistant Doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: The Key to Emotional Balance
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: The Key to Emotional Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The Key to Emotional Balance (KBA) program consists of eight sessions, each lasting 40-50 minutes, and aims to help participants develop emotional balance. The first session introduces the individual, introduces group rules, provides information about the program, and supports the client in identifying and expressing their emotions. The second session encourages the client to assess their energy-time intensity in their current and future balance models and, if deviations occur, to restructure them. The third session will help participants recognize their abilities in coping with bipolar illness and its symptoms and to use these abilities effectively. They will also be encouraged to identify factors that hinder their ability to use their abilities and focus on their developed abilities. The fourth session will focus on developing a "positive" perspective, enabling them to approach bipolar illness and its symptoms from a positive perspective. The fifth session will support participants
  Interventions: Behavioral: The Key to Emotional Balance
- Control (No Intervention): After an explanation of the study is provided to the individuals in the control group, verbal and written consent will be obtained from those who agree to participate in the study. Individuals who agree to participate will be administered an "Introductory Information Form," the "Difficulties in Emotion Regulation," the "Recovery Assessment Scale," and the Life Goals Scale in the Context of Positive Psychotherapy. Patients in this group will not receive any treatment other than their routine treatment. At the end of the study, individuals will be administered the "Difficulties in Emotion Regulation," the "Recovery Assessment Scale," and the Life Goals Scale in the Context of Positive Psychotherapy. Subsequently, the individuals in the control group will undergo all of the same sessions.

INTERVENTIONS:
Behavioral: The Key to Emotional Balance — The Key to Emotional Balance (KBA) program consists of eight sessions, each lasting 40-50 minutes, and aims to help participants develop emotional balance. The first session introduces the individual, introduces group rules, provides information about the program, and supports the client in identifying and expressing their emotions. The second session encourages the client to assess their energy-time intensity in their current and future balance models and, if deviations occur, to restructure them. The third session will help participants recognize their abilities in coping with bipolar illness and its symptoms and to use these abilities effectively. They will also be encouraged to identify factors that hinder their ability to use their abilities and focus on their developed abilities. The fourth session will focus on developing a "positive" perspective, enabling them to approach bipolar illness and its symptoms from a positive perspective. The fifth session will support participants
  Arms: Experimental

SUMMARY:
This randomized controlled experimental study aimed to evaluate the effects of the Key to Emotional Balance (KBA) psychoeducational program, based on the Balance Model of Positive Psychotherapy (PPT), on indicators of emotion regulation difficulties, recovery, and purpose in life in adults with bipolar disorder. Intervention and control groups (n=37 each; total n=74) will be formed through simple random assignment. The intervention will consist of eight individual sessions, each lasting 40-50 minutes. Data will be collected using the Difficulty in Emotion Regulation, Recovery Assessment Scale, and the Life Goals Scale in the Context of PPT. Measurements will be conducted as a pretest and posttest.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of bipolar I or bipolar II disorder according to the DSM-5.
2. Being between 18 and 65 years of age.
3. Being literate and having the cognitive capacity to participate in written questionnaires.
4. Being in a stable mood/remission (neither severely manic nor severely depressed) at the start of the study.
5. Being on medication or willing and able to comply with treatment.
6. Voluntarily agreeing to participate in the study and signing the informed consent form.

Exclusion Criteria:

1. Being in an episode of acute mania or severe depression.
2. Having a diagnosis of another serious psychiatric disorder such as schizophrenia, schizoaffective disorder, severe anxiety disorder, or obsessive-compulsive disorder (OCD).
3. Cognitive impairments, such as dementia, severe cognitive impairment, or mental retardation, that would prevent participation in the recommended therapy.
4. Individuals with a history of substance abuse within the last 6 months or ongoing active substance use.
5. Individuals who have attempted suicide within the last 6 months or who currently have suicidal thoughts (patients at high risk of suicide).
6. Refusal to attend regular therapy sessions or severe resistance to psychotherapy.
7. Individuals who are not compliant with recommended medication for bipolar disorder.
8. Serious medical problems or chronic conditions that would prevent recommended psychotherapy (e.g., uncontrolled epilepsy or serious cardiovascular disease).
9. Inability to speak Turkish sufficiently to understand the questionnaires and therapeutic interventions or difficulty communicating.

Exclusion Criteria:

1. Not attending psychoeducation sessions more than three times or not completing any of the pretest and posttest measures of the data collection forms.
2. Relapse of disease during the study and inability to comply with the program.
3. Participating in any other program while the study is ongoing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Difficulty in Emotion Regulation | Timeframe: Pre-test, 8 weeks later
  The short form of the scale was developed by Bjureberg and colleagues (2016). The scale is a 5-point Likert-type scale consisting of 16 items. It includes five subscales. These are: difficulty in making sense of emotions when experiencing negative emotions (clarity), difficulty in performing goal-directed behaviors when experiencing negative emotions (goals), difficulty in applying emotion regulation strategies when experiencing negative emotions (strategies), difficulty in accepting negative emotions (non-acceptance), and difficulty in maintaining impulse control when experiencing negative emotions (drive). The validity and reliability study of the scale, which consists of the sub-dimensions of goals (questions 3, 7, 15), strategies (questions 5, 6, 12, 14, 16), non-acceptance (questions 9, 10, 13, openness (questions 1, 2) and impulse (questions 4, 8, 11), was carried out by Yiğit and Güzey-Yiğit (2017) in our country. It is observed that the Cronbach's Alpha internal consistency co

SECONDARY OUTCOMES:
Recovery Assessment Scale: | Timeframe: Pre-test, 8 weeks later
  The scale was developed by Corrigan and colleagues (2004) to measure various sub-dimensions of recovery from the perspective of individuals diagnosed with mental illness and adapted to Turkish by Güler and Gurkan (2019). The scale consists of 24 items and 5 sub-dimensions. It is a 5-point Likert-type scale. The sub-dimensions of the scale include: self-confidence and hope sub-dimension: items 7, 8, 9, 10, 11, 12, 13, 14, and 21; help-seeking behavior sub-dimension: items 18, 19, and 20; goal and achievement orientation sub-dimension: items 1, 2, 3, 4, and 5; trust in others sub-dimension: items 6, 22, 23, and 24; and coping with symptoms sub-dimension: items 15, 16, and 17. There are no reverse items in the scale. Possible scores range from 24 to 120. The total scale score is the sum of the scores obtained from each item. While there is no cutoff score, it is assumed that improvement scores increase as the total scale score increases. Cronbach's alpha values for the scale subscales
Determining Life Goals in the Context of Positive Psychotherapy (PPBYABÖ): | Timeframe: Pre-test, 8 weeks later
  This scale was developed by Eryılmaz (2012). It measures whether individuals have determined their life goals in three areas. The scale is a nine-item, four-point Likert-type scale with three subdimensions: achievement (career) goals, relationship goals, and body (sense) goals. The Body Goals dimension of the scale includes individuals' goals related to physical relaxation; the Relationship Goals dimension includes individuals' goals such as determining the characteristics of their future spouses and having children. The Success Goals dimension includes individuals' career goals. Items 1, 2, and 3 are related to achievement (career) goals; items 4, 5, and 6 are related to relationship goals; and items 7, 8, and 9 are related to body (sense) goals. The lowest score possible on the scale is 9, and the highest score is 36. The Cronbach Alpha value of the achievement (career) goals sub-dimension of the scale is 0.85, the Cronbach Alpha value of the relationship goals dimension is 0.73, an

IPD SHARING:
Plan to Share IPD: No